CLINICAL TRIAL: NCT05835219
Title: REBYOTA™ for the Prevention of Recurrence of Clostridioides Difficile Infection (CDI) in Adult Patients: An Observational Study
Brief Title: REBYOTA™ Prospective Registry
Acronym: ROAR
Status: Completed | Type: Observational
Sponsor: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Other Study IDs: 000422
Record Dates: First submitted 2023-04-18; First posted 2023-04-28 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Recurrence of Clostridium Difficile Infection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- REBYOTA™
  Interventions: Drug: REBYOTA™

INTERVENTIONS:
Drug: REBYOTA™ — REBYOTA™ is administered in the rectum

SUMMARY:
This is a prospective observational cohort study designed to collect data on patients who received REBYOTA™ for the prevention of rCDI in the routine care setting. As all data collected for this study are observational, the decision to prescribe REBYOTA™ is at the treating physician's discretion and independent from the decision to enroll the patient in the study. Data will be collected from patients' medical records after obtaining informed consent. Data about clinical history, CDI events (primary and recurrent: severity, treatment), CDI-related symptoms, treatments, medical procedures, Adverse Events(AEs), and healthcare resource utilization (i.e., hospitalizations and re-admissions) will be collected through 6 months of follow-up from the date of REBYOTA™ administration.

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent form (ICF)
* Age ≥ 18 years
* Diagnosis of rCDI as determined by the treating physician
* Completed antibiotic treatment for the presenting rCDI episode
* Prescription for REBYOTA™ to prevent rCDI according to the approved indication

Exclusion Criteria:

* Currently enrolled in an interventional clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects who have received antibiotic treatment for Clostridioides Difficile Infection
Sampling Method: Non-Probability Sample
Enrollment: 145 (Actual)
Dates: Start 2023-06-19 (Actual); Primary Completion 2025-08-29 (Actual); Study Completion 2025-08-29 (Actual)

PRIMARY OUTCOMES:
Proportion of patients without Recurrence of Clostridioides Difficile Infection (rCDI) (as determined by the treating physician) | 8 weeks after initial REBYOTA™ treatment

SECONDARY OUTCOMES:
Proportion of patients with sustained clinical response, defined as treatment success of the presenting rCDI episode and no new CDI episodes occurring for more than 8 weeks through 6 months after initial REBYOTA™ treatment | 6 months after initial REBYOTA™ treatment
Total number of CDI episodes | 6 months after initial REBYOTA™ treatment
Time to any CDI episode | 6 months after initial REBYOTA™ treatment
Daily mean changes in Clostridium difficile Infection-Daily Symptoms (CDIDaySyms™) scores from baseline to 7 days after REBYOTA™ administration | 7 days after REBYOTA™ administration
Hospitalizations and re-admissions during follow-up for up to 6 months (all-cause and CDI-related) after receiving REBYOTA™ | Up to 6 months after receiving REBYOTA™

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Compliance, Study Director — Ferring Pharmaceuticals
Locations (39):
- United States (39):
  - Ferring Investigational Site, Chandler, Arizona
  - Ferring Investigational Site, Chula Vista, California
  - Ferring Investigational Site, Murrieta, California
  - Ferring Investigational Site, Oceanside, California
  - Ferring Investigational Site, Sacramento, California
  - Ferring Investigational Site, Hamden, Connecticut
  - Ferring Investigational Site, Gainesville, Florida
  - Ferring Investigational Site, Orlando, Florida
  - Ferring Investigational Site, Port Orange, Florida
  - Ferring Investigational Site, Tampa, Florida
  - Ferring Investigational Site, Zephyrhills, Florida
  - Ferrin Investigational Site, Atlanta, Georgia
  - Ferring Investigational Site, La Grange, Georgia
  - Ferring Investigational Site, Savannah, Georgia
  - Ferring Investigational Site, Burr Ridge, Illinois
  - Ferring Investigational Site, Maywood, Illinois
  - Ferring Investigational Site, Iowa City, Iowa
  - Ferring Investigational Site, Wichita, Kansas
  - Ferring Investigational Site, Jefferson, Louisiana
  - Ferring Investigational Site, Boston, Massachusetts
  - Ferring Investigational Site, Worcester, Massachusetts
  - Ferring Investigational Site, Detroit, Michigan
  - Ferring Investigational Site, Farmington Hills, Michigan
  - Ferring Investigational Site, Omaha, Nebraska
  - Ferring Investigational Site, Teaneck, New Jersey
  - Ferring Investigational Site, New York, New York
  - Ferring Investigational Site, Rochester, New York
  - Ferring Investigational Site, Stony Brook, New York
  - Ferring Investigational Site, Fargo, North Dakota
  - Ferring Investigational Site, Cincinnati, Ohio
  - Ferring Investigational Site, Middleburg Heights, Ohio
  - Ferring Investigational Site, DuBois, Pennsylvania
  - Ferring Investigational Site, Pittsburgh, Pennsylvania
  - Ferring Investigational Site, Charleston, South Carolina
  - Ferring Investigational Site, Knoxville, Tennessee
  - Ferring Investigational Site, Dallas, Texas
  - Ferring Investigational Site, Houston, Texas
  - Ferring Investigational Site, West Jordan, Utah
  - Ferring Investigational Site, Charlottesville, Virginia

IPD SHARING:
Plan to Share IPD: No